CLINICAL TRIAL: NCT01086059
Title: Humira (Adalimumab) Pregnancy Exposure Registry: OTIS Rheumatoid Arthritis in Pregnancy Project
Brief Title: OTIS Humira Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: The Organization of Teratology Information Specialists (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Christina Chambers, Principal Investigator, Professor Department of Pediatrics, University of California, San Diego
Other Study IDs: M03-604
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2021-04

CONDITIONS: Crohn's Disease; Rheumatoid Arthritis
Keywords: Autoimmune diseases; adalimumab; pregnancy; birth defects; TNF; Tumor necrosis factor
MeSH Terms: conditions — Crohn Disease; Arthritis, Rheumatoid; Autoimmune Diseases; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Cohort 1 - Exposure cohort: Pregnant women with a current diagnosis of RA, JRA, or Crohn's disease who have used adalimumab in the first trimester of pregnancy for any length of time from the date of conception.
- Cohort 2 - Matched Diseased Comparison Cohort: Pregnant women with a current diagnosis of RA, JRA, or Crohn's disease who have not used adalimumab or any TNF antagonist in pregnancy.
- Cohort 3-Non-Diseased Comparison Cohort: Pregnant women without a current diagnosis of an autoimmune disease and who have not used adalimumab or any TNF antagonist at any time in pregnancy nor have they been exposed to any known human teratogen during pregnancy.
- Cohort 4 - Registry Group: Pregnant women who have used adalimumab for any length of time following the first day of the last menstrual period until the end of pregnancy who do not meet Cohort 1 inclusionary criteria.

SUMMARY:
The purpose of the OTIS Autoimmune disease in pregnancy study is to monitor planned and unplanned pregnancies exposed to certain medications, to evaluate the possible teratogenic effect of these medications and to follow live born infants for one year after birth. With respect to fetal outcome, it is important to evaluate the spectrum of outcomes that may be relevant to a medication exposure during pregnancy, and these include both easily recognizable defects that are visible at birth, as well as, more subtle or delayed defects that may not be readily identifiable without special expertise and observation beyond the newborn period.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who reside in the United States, Canada or Puerto Rico.
Sampling Method: Non-Probability Sample
Enrollment: 944 (Actual)
Dates: Start 2003-11; Primary Completion 2016-08 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Major malformations | Throughout pregnancy and up to 1 year of life
  The primary objective of the study is to evaluate the effect of certain medications when used in the first trimester of pregnancy with respect to major structural birth defects of newborns.

SECONDARY OUTCOMES:
Minor malformations | At dysmorphological exam
  One secondary objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to potential minor malformations.
Pregnancy outcome | Throughout pregnancy
  Another objective of the study is to evaluate the effects of certain medications when used during pregnancy with respect to spontaneous abortion, stillbirth, and preterm delivery.
Infant follow-up | Throughout pregnancy and up to 1 year of life
  Pre- and post-natal fetal and infant growth, health and development

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Jones, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Chambers CD, Johnson DL, Xu R, Luo Y, Lopez-Jimenez J, Adam MP, Braddock SR, Robinson LK, Vaux K, Lyons Jones K; OTIS Collaborative Research Group. Birth outcomes in women who have taken adalimumab in pregnancy: A prospective cohort study. PLoS One. 2019 Oct 18;14(10):e0223603. doi: 10.1371/journal.pone.0223603. eCollection 2019. PMID 31626646
- See also: Official Research Website of the Organization of Teratology Information Specialists, Studies Coordinated at the University of California, San Diego — https://mothertobaby.org/pregnancy-studies/